CLINICAL TRIAL: NCT01295931
Title: Diagnostic Nodal Staging for Melanoma With Nuclear and Near-Infrared (NIR) Molecular Optical Imaging
Brief Title: Nuclear and Near-Infrared (NIR) Imaging in Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-0577; U54CA136404 (NIH)
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Melanoma
Keywords: Near-infrared; NIR; Indocyanine green; ICG; Melanoma; Fluorescent dyes; Lymph nodes; Experimental camera
MeSH Terms: conditions — Melanoma | interventions — Indocyanine Green; X-Rays; Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IC-Green + Imaging (Experimental): Indocyanine Green (IC-Green) Injections + Imaging
  Interventions: Drug: Indocyanine Green (IC-Green); Procedure: Imaging

INTERVENTIONS:
Drug: Indocyanine Green (IC-Green) — 5 intradermal injections, 25 µg IC-Green in 0.1 mL of saline, in locations on the extremity (i.e. arm or leg) correlating with the tumor draining nodal basin to begin. Corresponding injections performed on the contralateral limbs.
  Other Names: ICG
Procedure: Imaging — Nonradioactive optical imaging with indocyanine green as a fluorescent contrast agent prior to sentinel lymph node biopsy or lymph node surgery.
  Other Names: near-infrared; NIR; NIR fluorescence imaging

SUMMARY:
Objectives:

1. To determine the feasibility of using microdose amounts of near-infrared (NIR) fluorescent contrast agent to image tumor-draining and contralateral lymphatics in melanoma patients prior to standard-of-care sentinel lymph node biopsy OR completion lymph node dissection (axillary or inguinofemoral)
2. To determine the feasibility of using nonradioactive optical imaging techniques with indocyanine green (ICG) as a fluorescent contrast agent to characterize lymphatic architecture and function by correlating the observed lymphatic structure and function with tumor and nodal status as determined from standard-of-care immunohistochemical evaluation.

DETAILED DESCRIPTION:
Indocyanine Green Injections:

IC-Green Injections:

If you are found to be eligible to take part in this study, you will receive a total of 10-16 injections of IC-Green through a needle in your arms or legs, starting in your hands or feet (5-8 on each arm/leg), depending on the location of the tumor. You may receive additional injections in the torso, if there is a tumor in the torso area and the study doctor thinks it is needed. The study doctor will discuss the number of injections that you will receive in more detail. The injections will be given to you before surgery and all injections will be given intradermally (into or between layers of the skin).

The IC-Green injections will allow researchers to see how fluid flows through your body during imaging. This information may help future researchers more easily locate lymph nodes in patients scheduled for lymph node surgery.

After all of the IC-Green injections have been given, the imaging procedure will begin. To perform the imaging procedures, researchers will use an experimental camera that shines a special red light onto your skin causing the IC-Green to glow when the images are taken. The red light is like the red light in a grocery store scanner. The imaging procedure will take about 1 hour to complete and will be performed before and during the surgery.

Before the IC-Green injections and again during the imaging procedure, a member of the research staff will monitor and record your vital signs (blood pressure, breathing rate, heart rate, and temperature). Vital sign measurements will be taken every 15 minutes for 1 hour after the IC-Green injections, and every 30 minutes during the second hour. A study staff member will also closely monitor the injection site at these times for possible side effects. A study staff member will call you the next day and ask you to take your temperature. This phone call should last about 10 minutes.

Length of Study:

After all of the images have been taken, and the follow-up evaluation is complete, your participation in this study will be over.

Follow-Up Evaluation:

If you spend the night in the hospital after surgery, a study staff member will visit you in person the day after surgery. At this visit, your temperature will be recorded, you will be asked how you are feeling, and if you have experienced any side effects. The visit should last about 10 minutes.

If you do not spend the night in the hospital after surgery, you will be contacted by phone the day after the surgery and you will be asked what your current temperature is, how you are feeling, and if you have experienced any side effects. The phone call should last about 10 minutes.

This is an investigational study. IC-Green is FDA approved and commercially available for assessment of cardiac output, hepatic function, liver blood flow, ophthalmic angiography, and mapping heart, liver, and eye function. The use of IC-Green for mapping the lymph nodes in melanoma patients is investigational.

IC-Green is FDA approved to be injected into the vein. Giving IC-Green injections into or between layers of the skin and the device that is used to give the injections are investigational. The experimental camera, and the images taken with it, are being used for research purposes only and will not be used to manage your treatment.

Up to 18 patients will take part in Part 1 of this study. All will be enrolled at MD Anderson.

Complete Lymph Node Dissection:

If you agree to participate in this part of the study, you will have additional imaging performed before the surgery and again in your follow-up visit.

The imaging will be performed at MD Anderson just before the surgery and during your regularly scheduled standard of care follow-up visit about 4-6 months after surgery to learn what the lymphatic channels look like after completely healing from surgery.

Before each imaging session, you will receive a total of 10-16 injections of IC-Green through a needle in your arms and hands or legs and feet, (5-8 on each arm/leg), depending on the location of the tumor. Researchers will use the experimental camera to perform the imaging procedure. You may receive additional injections in the torso, if there is a tumor in the torso area and the study doctor thinks it is needed.

The imaging procedures will take up to 2 hours to complete each time.

For all participants, before the IC-Green injections and again during the imaging procedure, a member of the research staff will monitor and record your vital signs (blood pressure, breathing rate, heart rate, and temperature). Vital sign measurements will be taken every 15 minutes for 1 hour after the IC-Green injections, and every 30 minutes during the second hour. A study staff member will also closely monitor the injection site at these times for possible side effects.

Length of Study:

Your participation will be over after all the images have been taken and the long-term follow-up is complete.

This is an investigational study. IC-Green is FDA approved and commercially available for assessment of cardiac output, hepatic function, liver blood flow, ophthalmic angiography, and mapping heart, liver, and eye function. The use of IC-Green for mapping the lymph nodes in melanoma patients is investigational.

IC-Green is FDA approved to be injected into the vein. Giving IC-Green injections into or between layers of the skin and the device that is used to give the injections are investigational. The experimental camera, and the images taken with it, are being used for research purposes only and will not be used to manage your treatment.

Up to 6 patients will participate in this part of the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older
2. Diagnosis of invasive melanoma with (ARM A) biopsy documenting a T2 (greater than 1 mm thickness) primary tumor undergoing standard of care sentinel lymph node biopsy (SLN) for definitive pathologic staging, OR (ARM B) documented node-positive (stage III) disease undergoing standard-of-care axillary or inguinofemoral lymph node dissection for regional disease control.
3. Negative urine pregnancy test within 72 hours prior to study drug administration, if female of childbearing potential.
4. Female of childbearing potential who agrees to use a medically accepted method of contraception for a period of one (1) month following the study. Medically acceptable contraceptives include (i) hormonal contraceptives such as birth control pills, Depo-Provera, or Lupron Depot) if such is approved by the subject's Oncologist; (ii) barrier methods (such as a condom or diaphragm used with a spermicide, or (iii) an intrauterine device (IUD). Non-childbearing potential is defined as physiologically incapable of becoming pregnant, including any female who is post-menopausal; postmenopausal is defined as the time after which a woman has experienced 12 consecutive months of amenorrhea (lack of menstruation).
5. For patients undergoing a complete axillary or inguinofemoral lymph node dissection a positive previous sentinel lymph node or a positive fine needle aspirate or core biopsy of their axillary or inguinofemoral lymph nodes.

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Persons who are allergic to iodine
3. A female of child-bearing potential who does not agree to use an approved contraceptive for one month after study participation.
4. History of ipsilateral axillary or femoral surgery not including previous sentinel lymph node biopsy procedure.
5. Persons who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Nodes Identified by Indocyanine Green (ICG) Among All Resected Lymph Nodes | 18-24 hours after procedure
  Procedure feasible if 18 out of 24 evaluable patients have 80% or more nodes identified by ICG among all resected nodes. Descriptive analyses performed to report the mean percentage and its 95% confidence interval of the nodes identified by ICG among the total resected nodes of all evaluable subjects. Outcome will be tabulated by age, different tumor stage, nodal status, and body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Janice N. Cormier, MD, MPH, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org